CLINICAL TRIAL: NCT01666132
Title: METHOD - Phase I/II Study of Intramyocardial Injection of Bone Marrow Derived Mononuclear Cells in Chronic Ischemic Disease
Brief Title: METHOD - Bone Marrow Derived Mononuclear Cells in Chronic Ischemic Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the slow recruitment process and the progress of newer cell types we decided to stop the trial after the phase 1 (after 10 patients included)
Sponsor: Cardiocentro Ticino (Other)
Responsible Party: Principal Investigator, Daniel Suerder, MD; senior attendant of Cardiology, Cardiocentro Ticino
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: METHOD
Record Dates: First submitted 2011-06-27; First posted 2012-08-16 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Ischemic Heart Disease
Keywords: LVEF < 40%

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intramyocardial injection of BM cells (Experimental)
  Interventions: Other: intramyocardial injection of BM cells
- Intramyocardial / intracoronary injection of BM cells (Experimental)
  Interventions: Other: intramyocardial / intracoronary injection of BM cells
- control (Other)
  Interventions: Other: Best medical therapy

INTERVENTIONS:
Other: intramyocardial injection of BM cells — only intramyocardial, NOGA guided injection on BM cells.
  Arms: Intramyocardial injection of BM cells
Other: intramyocardial / intracoronary injection of BM cells — combination of intramyocardial, NOGA guided injection of BM cells and intracoronary injection of those cells
  Arms: Intramyocardial / intracoronary injection of BM cells
Other: Best medical therapy — initially no intervention; crossover to therapy 6 months after enrollment
  Arms: control

SUMMARY:
Intramyocardial, NOGA guided injection of bone marrow derived mononuclear cells in patients with chronic ischemic heart disease and LVEF < 40%. The primary objective is to determine whether the administration of the cells improves recovery of the left ventricular function. Secondary objective is the finding of clinical or paraclinical parameters to predict potential benefits of the treatment (basing on MRI characteristics such as size, transmurality of the myocardial infarction and peri-lesional ischemia).

In the first part of the study 10 patients are treated without control group. This phase serves as feasibility and safety part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic cardiac ischemic disease at least 4 months after one ore more myocardial infarctions in a stable phase of the disease without option for revascularization
* LVEF at echocardiography ≤ 40%
* Significant regional LV wall motion dysfunction in the infarct related territory
* Symptoms NYHA II-IV or CCS II-III (at least class III according to one of the two classifications)
* Patient agrees to comply with all follow-up evaluations
* Age > 18 years old
* Patient has been informed of the nature of the clinical trial and agrees to its provision and has provided written informed consent

Exclusion Criteria:

* Abnormal regional wall motion outside the infarct region
* Need for revascularization in a non infarct-related coronary within 6 months
* Patient has moderate to severe aortic valve disease, aortic or mitral prosthetic valve
* Patient has a significant mitral valve insufficiency (Effective Regurgitant office - ERO - > 0.2 cm2 with possibility of mitral valve surgery
* Left ventricular thrombus at echocardiography
* LV-aneurysma planned surgical aneurysmectomy
* LV-wall thickness < 5mm in the target territory
* Congenital heart disorder of hemodynamic relevance
* Known active infection or chronic infection with HIV, HBV or HCV
* Chronic inflammatory disease
* Serious concomitant disease with a life expectancy of less than one year
* Follow up impossible (no fixed abode, etc)
* Contraindication for cardiac MRI (i.e. pace maker, neurostimulator, claustrophobia)
* Severe renal failure (creatinine > 250 mmol/l)
* Relevant liver disease (GOT > 2x norm or spontaneous INR > 1,5)
* Anemia (Hb < 8.5 mg/dl), Thrombocytopenia (< 100.000/µl)
* Women of child bearing potential or pregnancy
* Participation at a clinical trial in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Troponin samples | 1 day after cell injection
  Measurements of Troponine after cell injection
Number of patients with adverse events at short term | within 1 week after cell injection
Number of patients with adverse events at mid/long term | up to 12 months after cell injection

SECONDARY OUTCOMES:
change in LVEF | 6 months vs. baseline
  First 10 patients + following randomization phase (n = 54); assessment of short term safety (1 week), Adverse events within 1 year; efficacy measurements 6 months after treatment
change in Quality of life | 6 months vs. baseline
change in Vo2 max | 6 months vs. bl
  change in functional status (Vo2 max)

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiocentro Ticino, Lugano, Switzerland

REFERENCES:
- [Derived] Maffessanti F, Prinzen FW, Conte G, Regoli F, Caputo ML, Suerder D, Moccetti T, Faletra F, Krause R, Auricchio A. Integrated Assessment of Left Ventricular Electrical Activation and Myocardial Strain Mapping in Heart Failure Patients: A Holistic Diagnostic Approach for Endocardial Cardiac Resynchronization Therapy, Ablation of Ventricular Tachycardia, and Biological Therapy. JACC Clin Electrophysiol. 2018 Jan;4(1):138-146. doi: 10.1016/j.jacep.2017.08.011. Epub 2017 Nov 6. PMID 29600778
- [Derived] Surder D, Radrizzani M, Turchetto L, Cicero VL, Soncin S, Muzzarelli S, Auricchio A, Moccetti T. Combined delivery of bone marrow-derived mononuclear cells in chronic ischemic heart disease: rationale and study design. Clin Cardiol. 2013 Aug;36(8):435-41. doi: 10.1002/clc.22148. Epub 2013 May 29. PMID 23720276